CLINICAL TRIAL: NCT06785142
Title: The Effects of a Multi-ingredient 'relaxation' Shot on Mood At Rest and During a Laboratory Stressor in Healthy Adults: a Randomized, Double-blind, Placebo-controlled, Crossover Trial
Brief Title: Investigation of a Dietary Supplement Liquid Shot Product on Aspects of Mood Both At Rest and During a Laboratory Stressor Task.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Water Street Collective (Industry)
Collaborators: HCD Research (Industry); British American Tobacco (Investments) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: HCD J8880
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Mood; Stress; Alertness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- AABB (Other): The order of study product to be consumed over 4 session will be: Placebo, Placebo, Experimental, Experimental
  Interventions: Dietary Supplement: Functional Shot; Dietary Supplement: Placebo Shot
- ABBA (Other): The order of study product to be consumed over 4 session will be: Placebo, Experimental, Experimental, Placebo
  Interventions: Dietary Supplement: Functional Shot; Dietary Supplement: Placebo Shot
- BAAB (Other): The order of study product to be consumed over 4 session will be: Experimental, Placebo, Placebo, Experimental
  Interventions: Dietary Supplement: Functional Shot; Dietary Supplement: Placebo Shot
- BBAA (Other): The order of study product to be consumed over 4 session will be: Experimental, Experimental, Placebo, Placebo
  Interventions: Dietary Supplement: Functional Shot; Dietary Supplement: Placebo Shot

INTERVENTIONS:
Dietary Supplement: Functional Shot — 60ml functional energy shot contained a proprietary blend of L-theanine, chamomile, lemon balm, ginseng and vitamins
Dietary Supplement: Placebo Shot — Placebo 60 ml Shot, matched in volume, taste and colour and but did not contain any active ingredients

SUMMARY:
This is a single center, randomized, double blind, placebo-controlled, crossover study to determine the acute effect of a developmental dietary supplement liquid shot product of aspect of mood both at rest and during laboratory stressor task. The study will be conducted in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participants that, on average, consume less than 400 mgs of caffeine per day and less than 14 units of alcohol per week.
2. Participants that are in good physical and mental health.
3. Participants that are willing to come in-person to participate in the research.
4. Participants that are able to provide written informed consent to participate in the study and will have agreed to abide by the study restrictions, requirements and protocol.
5. Participants must, in the opinion of the Principal Investigator (or designee), demonstrate the ability to comprehend the informed consent form (ICF), be able to communicate well with the Investigator, understand and comply with the requirements of the study, and be judged suitable for the study.
6. Participants must be available to complete the study.
7. Participants must be willing to fast from food/beverages (other than water) for at least one hour prior to each session, from caffeine for at least three hours prior and from alcohol for at least twelve hours prior.

Exclusion Criteria:

1. Participants that are not UK citizens or residents.
2. Participants that have a medical condition, including but not limited to heartbeat/rhythm irregularities, past heart attacks, been diagnosed with heart disease, seizure disorder, liver condition, blood clotting disorder, endocrine-related medical diagnosis (such as diabetes, thyroid, etc.), asthma/emphysema/COPD, serious health condition (i.e., cancer, etc.), blindness, insomnia, narcolepsy, anxiety, depression, hypertension, or deafness. If a participant has any other medical condition or metabolic condition that prevents them from being able to fast for one hour, they will not be allowed to participate in this study.
3. Participants likely to be experiencing fluctuations in mood state such as those that have recently had surgery, changed jobs, experienced the death of a close friend/family member, or are in the process of getting divorced.
4. Participants that do not sleep during the night, do not work day-shift hours, or have other factors that impact their sleep schedule such as an inconsistent work schedule, or having disruptions in their sleep due to being the caretaker of a child/adult, dealing with chronic pain or having a sleep disorder (such as Narcolepsy, Insomnia, or Sleep Apnoea).
5. Participants that have a loss of taste or smell or are currently suffering from a virus/infection that affects their ability to taste or smell.
6. Participants that currently or in the past have been diagnosed with a chronic cold or sinus condition.
7. Participants that have paralysis which effects the upper body, or are colour-blind, as this could impact their ability to complete the tasks in the study.
8. Participants that use recreational drugs or that are currently taking medication (except for a contraceptive), or other drugs including non-prescription (over the counter) medications, non-prescription painkillers such as paracetamol (acetaminophen), ibuprofen or aspirin.
9. Participants that are pregnant, breastfeeding (or pumping/expressing) or intend to become pregnant within the next six months.
10. Participants that currently use cannabinoid products, smoke cigarettes or use any tobacco or nicotine products.
11. Participants that are allergic or sensitive to any of the product ingredients.
12. Participants that have experienced or that have members of their household that have experienced any of the following symptoms in the past 14 days: cough, shortness of breath or difficulty breathing, fever, chills, repeated shaking with chills (rigors), sore throat, or new loss of taste or smell.
13. Participants that have tested positive, or have been in contact with, someone who has tested positive for Coronavirus/COVID-19 in the past 14 days.
14. Participants that are currently or have participated in market research in the last 30 days.
15. Participants that currently work (or who have an immediate family member who works) for a market research, marketing, advertising, public relations, pharmaceutical, food/beverage or tobacco company.
16. Participants who cannot satisfactorily complete the training/Familiarisation Session with the Investigational Products and the relevant assessments.
17. Participants who are unwilling or unable to comply with the study requirements and restrictions including those outlined in the Participant Handbook.

Ages: 29 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-01-14 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the State-Trait Anxiety Inventory up to 135 minutes for the functional shot versus placebo shot. | From Baseline to 135 minutes post trial product consumption
  The STAI 'State' subscale contains 6 statements each responded to with a 4-point Likert scale. Scores range from 6-24, where higher scores indicate higher anxiety.

SECONDARY OUTCOMES:
Change from Baseline in Mood via Visual Analogue Mood Scales (VAMS) up to 135 minutes for the functional shot versus placebo shot. | From Baseline to 135 minutes post trial product consumption
  Comprising of 18 visual analogue scales anchored by pairs of antonymic mood/state adjectives (e.g. Alert - Inattentive; Lethargic - Energetic) on 0-100% line. The individual item scores are combined to give an average (% along the line) score on three factors that had previously been derived by factor analysis: 'Alertness', 'Tranquility' and 'Stress'. Higher scores indicate a higher level of each factor.
Change from Baseline in Mood via Visual Analogue Scales (VAS) up to 135 minutes for the functional shot versus placebo shot. | From Baseline to 135 minutes post trial product consumption
  0-100 mm subjective rating scale from none to strongest feelings, for clam, sleepy, nervous and in control. Higher scores indicate a higher level of each factor.
Change from Baseline in physiological state via POMS up to 135 minutes for the functional shot versus placebo shot. | From Baseline to 135 minutes post trial product consumption
  a 37-item inventory, the individual item scores of which are collapsed into six dimensions of mood: anger/hostility, confusion/bewilderment, depression/dejection, fatigue/inertia, tension/anxiety, and vigour/activity. Higher scores indicate a higher level of each factor.
Change from Baseline in physiological state via Self-Assessment Manikin up to 135 minutes for the functional shot versus placebo shot. | From Baseline to 135 minutes post trial product consumption
  The three single-item scales, each comprising nine simple line-drawn human figures with titrated emotional connotations, measure the participants current emotional position between happiness and sadness (Pleasure scale), relaxed and excited (Arousal scale), and feeling no-control to feeling in full-control (Dominance scale). Higher scores indicate a higher level of each factor.

CONTACTS AND LOCATIONS:
Locations (1):
- Sago London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided